CLINICAL TRIAL: NCT04275869
Title: Efficacy of an Internet-based Intervention to Promote a Healthy Lifestyle on the Reproductive Parameters of Overweight and Obese Women: a Randomised Controlled Trial
Brief Title: Internet-based Intervention to Promote a Healthy Lifestyle on the Reproductive Parameters of Overweight and Obese Women
Acronym: HLRP-RCT
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants enrolled
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital Universitario de la Plana (Other)
Responsible Party: Principal Investigator, Juan F. Lisón Párraga, Dr, Head of Medicine, Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UNIVERSITY CARDENAL HERRERA-25
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Infertility, Female
Keywords: infertility; obesity; physical activity; nutrition; internet
MeSH Terms: conditions — Obesity; Infertility, Female; Infertility; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Healthy Lifestyle (Experimental): A 3-month internet-based program focusing on the promotion of healthy lifestyles. The treatment protocol comprises 9 modules which incorporate psychological strategies to promote healthy lifestyles by gradually changing eating and physical activity habits.
  Interventions: Other: Healthy Lifestyle
- Control Group (No Intervention): Control group will receive the standard treatment which consists of regular gynaecological visits; the Reproduction Service gynaecologists will recommend healthy lifestyle habits and give the patients a document detailing a specific diet they should follow for weight loss.

INTERVENTIONS:
Other: Healthy Lifestyle — A 3-month internet-based program focusing on the promotion of healthy lifestyles. The treatment protocol comprises 9 modules which incorporate psychological strategies to promote healthy lifestyles by gradually changing eating and physical activity habits.
  Arms: Experimental Healthy Lifestyle

SUMMARY:
Obesity and overweight are among the problems that produce infertility. The combination of diet and exercise to achieve weight loss are currently considered an effective intervention for the improvement of reproductive parameters in overweight or obese infertile women.

Aim: to evaluate the effectiveness of an online program to promote a healthy lifestyle among women who are overweight or obese who also have a diagnosis of infertility and are on the waiting list for in vitro fertilisation treatment

DETAILED DESCRIPTION:
Weight management problems (being obese or overweight) are among the problems that produce infertility. The combination of diet and exercise to achieve weight loss are currently considered an effective intervention for the improvement of reproductive parameters in overweight or obese infertile women.

Aim: to evaluate the effectiveness of a 3-month internet-based program focusing on the promotion of healthy lifestyles (especially weight loss and healthy eating and physical exercise habits) in women who also have a diagnosis of infertility and are on the waiting list for IVF treatment.

Design: randomised controlled trial Setting: Hospital La Plana (Villarreal)

ELIGIBILITY:
Inclusion Criteria:

* women of childbearing age
* overweight (BMI > 25 kg/m2) or obese (BMI > 30 kg/m2)
* diagnosed with primary infertility -access to the internet-

Exclusion Criteria:

* over 40 years
* morbid or extreme obesity (BMI > 40 kg/m2)
* bilateral obstruction of the fallopian tubes
* endometriosis
* women whose partner has a severe male factor (oligoasthenoteratozoospermia).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 0 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Spontaneous clinical pregnancy rate | 12 months
  The primary outcome will be the spontaneous clinical pregnancy rate (pregnancy with ultrasound visualisation of the gestational sac at week 7 of pregnancy) and evolution (pregnancy with ultrasound visualisation of the gestational sac and a heartbeat after 20 weeks of gestation).

SECONDARY OUTCOMES:
Body mass index (BMI) | 12 months
  Weight (in kilograms) and height (in meters) will be combined to report BMI in kg/m^2.
Abdominal perimeter | 12 months
  It will be measured with a tape-measure at the level of the navel (without compressing the skin tissue) and after drawing in air following one deep inhalation and exhalation.
Mediterranean Diet Adherence | 12 months
  Mediterranean Diet Adherence Screener (MEDAS) questionnaire used in the PREDIMED trial. This questionnaire has been validated for the Spanish population and assesses adherence to the Mediterranean diet.
Physical activity level | 12 months
  This is a self-administered questionnaire comprising 7 items which collects information about the physical activity the surveyee has completed in 7 days prior to completing the test. The IPAQ-SF will be used to calculate the total number of minutes and days the person has engaged in physical activity by adding all physical activity category scores from the prior 7 days together. This data will be converted into metabolic equivalent of task minutes per week (MET-min/week), using the formula published by Ainsworth et al., to classify their physical activity levels as 'high' (> 1,500 MET-min/week), 'moderate' (600-1,500 MET-min/week), or 'low' (< 600 MET-min/week).

CONTACTS AND LOCATIONS:
Overall Officials: JUAN FRANCISCO L PÁRRAGA, PhD, Principal Investigator — Cardenal Herrera University
Locations (1):
- Hospital La Plana de Villarreal, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: Undecided